CLINICAL TRIAL: NCT01610700
Title: Double Blind, Randomised, Parallel Group, Placebo Controlled Trial of a Combination of THC and CBD in Patients With Multiple Sclerosis, Followed by an Open Label Assessment and Study Extension
Brief Title: An Investigation of Delta-9-tetrahydrocannabinol (THC) and Cannabidiol (CBD) in Multiple Sclerosis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWMS0001 Part A
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GW-1000-02 (Experimental): Active treatment
  Interventions: Drug: GW-1000-02
- Placebo (Placebo Comparator): Control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GW-1000-02 — Containing THC (27 mg/ml):CBD (25 mg/ml), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring. The maximum permitted dose of study medication was eight actuations (22 mg THC and 20 mg CBD) in any three hour period, and 48 actuations (130 mg THC and 120 mg CBD) in any 24 hour period.
  Other Names: Sativex
  Arms: GW-1000-02
Drug: Placebo — Each actuation of placebo delivered the excipients only.
  Arms: Placebo

SUMMARY:
A study to compare the efficacy of GW-1000-02 [named Sativex® in Canada and also named Sativex® Oromucosal Spray] with placebo in relieving five key symptoms of Multiple Sclerosis after six weeks of therapy.

DETAILED DESCRIPTION:
Eligible subjects entered a one to two week baseline period; followed by a six week double blind, randomised, parallel group comparison of GW-1000-02 with placebo, self-titrated to symptom resolution or maximum tolerated dose. Existing medication continued at a constant dose.

Primary efficacy comparisons were made between symptom scores recorded during baseline and scores recorded at the end of the parallel group period.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years.
* Multiple Sclerosis of any type.
* Stable Multiple Sclerosis symptomatology during the four weeks before study entry.
* Symptoms of the required severity (>50 mm on a 100 mm Visual Analogue Scale severity scale) in least one of the specified impairment categories; spasticity, muscle spasms, disturbed bladder control, neuropathic pain, limb tremor.
* A stable medication regime during the four weeks before study entry.
* Willing to abstain from cannabis or cannabinoids for at least seven days before study entry, and during the study.
* Agreed either to use effective contraception during the study and for three months thereafter, or had been surgically sterilised or, if female, were post-menopausal.
* Clinically acceptable laboratory results for pre-study screening.
* Willing and able to undertake and comply with all study requirements.
* Willing and able to read, consider and understand the subject information and consent form and give written informed consent. Subjects unable to read or to sign the document procedures were treated as detailed in the Declaration of Helsinki.
* Willing for their general practitioner, and consultant if appropriate, to be informed of study participation.
* Willing for their name to be notified to Home Office for participation in the study.

Exclusion Criteria:

* Known or strongly suspected to be abusing drugs, including alcohol.
* Not prepared to abstain from cannabis or cannabinoids during the study.
* Current or past addiction to cannabis.
* Known or suspected to have had an adverse reaction to cannabinoids causing psychosis or other severe psychiatric illness.
* History of any type of schizophrenia, any other psychotic illness, or other significant psychiatric illness or personality disorder other than depression associated with chronic illness.
* Received any drug containing levodopa (Sinemet®, Sinemet plus®, Levodopa®, L-dopa®, Madopar®, Benserazide®).
* Serious cardiovascular disorder including angina, uncontrolled hypertension, or an uncontrolled symptomatic cardiac arrhythmia.
* Significant renal or hepatic impairment as shown in medical history or indicated by laboratory results.
* History of epilepsy.
* Terminal illness or other condition in which placebo medication would be inappropriate.
* Pregnant, lactating or at risk of pregnancy.
* Participated in any other clinical research study during the 12 weeks before study entry.
* Planned hospital admission between study entry and Visit 6.
* Planned travel outside the UK between study entry and Visit 6.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2001-05; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rivermead Rehabilitation Centre, Oxford, United Kingdom

REFERENCES:
- [Result] Wade DT, Makela P, Robson P, House H, Bateman C. Do cannabis-based medicinal extracts have general or specific effects on symptoms in multiple sclerosis? A double-blind, randomized, placebo-controlled study on 160 patients. Mult Scler. 2004 Aug;10(4):434-41. doi: 10.1191/1352458504ms1082oa. PMID 15327042

RESULTS

PARTICIPANT FLOW:
Groups:
- GW-1000-02: Contains Δ9 tetrahydrocannabinol (THC), 27 mg/ml: cannabidiol (CBD), 25 mg/ml delivered in 100 microlitre actuations by a pump action oromucosal spray. Maximum permitted dose was284 actuations (THC 130 mg: CBD 120 mg) in 24 hours.
- Placebo: Contains no active drug but colourants and excipients. Maximum permitted dose was 48 actuations in 24 hours.
Period: Overall Study
Arm/Group | GW-1000-02 | Placebo
Started | 80 | 80
Completed | 77 | 77
Not Completed | 3 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — subject took one dose of street cannabis | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GW-1000-02 | Placebo | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 74 | 148
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.96 (9.36) | 50.42 (9.33) | 50.69 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 52 | 99
  Male | 33 | 28 | 61
Region of Enrollment [Number; unit: participants]
  United Kingdom | 80 | 80 | 160

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Composite Primary Impairment Visual Analogue Scale Score at the End of 6 Weeks of Treatment
Description: This was achieved by measuring the change from baseline after six weeks of therapy in the severity of the primary impairment, a composite score from one of five Multiple Sclerosis symptom categories that subjects nominated as their most severe symptom. The severity scores were recorded using a 100 mm Visual Analogue Scale, where 0 = no problem and 100 = very bad. A decrease in score indicates an improvement.
Time Frame: baseline and 6 weeks
Population: All subjects randomised who received at least one dose of study medication and had any on-treatment evaluable efficacy data recorded were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- GW-1000-02: Contains Δ9 tetrahydrocannabinol (THC), 27 mg/ml: cannabidiol (CBD), 25 mg/ml delivered in 100 microlitre actuations by a pump action oromucosal spray. Maximum permitted dose was 48 actuations (THC 130 mg: CBD 120 mg) in 24 hours.
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 79 | 77
units on a scale | -25.32 (23.42) | -19.32 (27.02)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change in the primary impairment was compared between treatment groups using analysis of covariance (ANCOVA) with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.124, ANCOVA; Estimated mean treatment difference = -5.93, 95% CI [-13.52 to 1.65]

2. Secondary Outcome: Change From Baseline in Spasticity Visual Analogue Scale Score at the End of 6 Weeks of Treatment
Description: Severity scores over the last 24 hours were recorded using a 100 mm Visual Analogue Scale on one nominated day each week. Scores ranged from 0 = no problem to 100 = very bad. A decrease in score indicates an improvement.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 71 | 65
units on a scale | -23.44 (21.59) | -15.98 (23.46)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change in the spasticity visual analogue scale score was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.062, ANCOVA; Estimated mean treatment difference = -7.10, 95% CI 2-sided [-14.56 to 0.37]

3. Secondary Outcome: Change From Baseline in Pain Visual Analogue Scale Score at the End of 6 Weeks of Treatment
Description: Severity scores were recorded using a 100 mm Visual Analogue Scale. Scores ranged from 0 = no problem to 100 = very bad. A decrease in score indicates an improvement.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 39 | 48
units on a scale | -15.62 (21.76) | -13.06 (29.52)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change in the pain visual analogue scale score was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.731, ANCOVA; Estimated mean treatment difference = -1.88, 95% CI 2-sided [-12.73 to 8.96]

4. Secondary Outcome: Change From Baseline in Muscle Spasm Visual Analogue Scale Score at the End of 6 Weeks of Treatment
Description: as for outcome 3
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 51 | 56
units on a scale | -24.15 (20.99) | -21.04 (25.08)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change in the muscle spasm visual analogue scale score was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.443, ANCOVA; Estimated mean treatment difference = -3.30, 95% CI 2-sided [-11.82 to 5.21]

5. Secondary Outcome: Change From Baseline in Tremor Visual Analogue Scale Score at the End of 6 Weeks of Treatment
Description: as for outcome 3
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | -21.40 (24.41) | -15.70 (25.44)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change in the tremor visual analogue scale score was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.311, ANCOVA; Estimated mean treatment difference = -6.85, 95% CI 2-sided [-20.31 to 6.60]

6. Secondary Outcome: Change From Baseline in Bladder Problems Visual Analogue Scale Score at the End of 6 Weeks of Treatment
Description: as for outcome 3
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 55 | 57
units on a scale | -28.10 (25.87) | -21.61 (25.61)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change in bladder problems visual analogue scale score was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.154, ANCOVA; Median Difference (Final Values) = -6.26, 95% CI 2-sided [-14.90 to 2.38], Standard Error of Mean 4.36

7. Secondary Outcome: Subject Global Opinion of Effect on Multiple Sclerosis at the End of Treatment
Description: A 7-point Likert-type scale was used, with the question: 'Please assess the status of your multiple sclerosis since entry into the study using the scale below' with the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse or very much worse". At Visit 2 (Baseline) patients wrote a brief description of their Multiple sclerosis which was used at end of treatment to aid their memory regarding their symptoms at study start. The number of subjects that considered their condition to be better or much better at the end of treatment is presented.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 79 | 77
participants | 32 | 21
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The proportion of subjects with better/much better assessments was compared between groups using a Fisher's Exact Test; Test type: Superiority or Other; p = 0.293, Fisher Exact; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.77 to 2.43]

8. Secondary Outcome: Change From Baseline in Modified Ashworth Scale Score at the End of Treatment
Description: All 20 muscle groups were assessed for spasticity (using a 1-5 scale): 1= no increase in muscle tone to 5= passive movement is difficult and affected part is rigid in flexion or extension. The score for all 20 muscle groups were added to give a total score out of 100; minimum score was 20. A decrease in score indicates an improvement in condition. As such, a negative value indicates an improvement in score from baseline.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 73 | 70
units on a scale | -0.38 (2.51) | -0.58 (2.04)

9. Secondary Outcome: Change From Baseline in the Mean Beck's Depression Inventory (BDI-II) Score at the End of Treatment
Description: This was a 21-question multiple choice self-report inventory. Subjects' responses to the 21 questions were assigned a score ranging from zero (good) to three (bad), indicating the severity of the symptom. The sum of all BDI-II question scores indicated the severity of depression; score range 0-63. A decrease in score indicates an improvement in condition. As such, a negative value indicates in improvement in score from baseline.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 78 | 77
units on a scale | -2.1 (5.59) | -2.9 (6.53)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline in the mean Beck's Depression Inventory score at the end of treatment was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.450, ANCOVA; Estimated mean treatment difference = 0.69, 95% CI 2-sided [-1.11 to 2.50]

10. Secondary Outcome: Change From Baseline in the Mean Fatigue Severity Scale Questionnaire Score at the End of Treatment
Description: The Fatigue Severity Scale is a nine-item questionnaire developed to assess the level of fatigue due to neurological disease, were each assessed on a 0-6 scale (0= no fatigue and 6= severe fatigue). As such a decreased score indicates improvement, and a negative value indicates and improvement from baseline.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 78 | 76
units on a scale | -0.30 (1.14) | -0.09 (0.97)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change baseline in the mean Fatigue Severity Scale Questionnaire score at the end of treatment was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.427, ANCOVA; Estimated mean treatment difference = -0.12, 95% CI 2-sided [-0.43 to 0.18]

11. Secondary Outcome: Change From Baseline in the Mean Rivermead Mobility Index Score at the End of Treatment
Description: The Rivermead Mobility Index is a measure of subject self-mobilisation and was developed to enable rehabilitation professionals to document the effect(s) of interventions. This consisted of 15 questions relating to the dexterity and/or mobility of the patient. Each question had a 'yes' / 'no' answer which was scored as yes=1 no=0. The summary parameter was the total for the 15 questions, with a maximum score of 15. An increased score indicates improvement. As such, a positive value indicates an improvement in score from baseline.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 79 | 77
units on a scale | 0.2 (1.68) | -0.0 (1.80)

12. Secondary Outcome: Change From Baseline in the Mean Total 28-item General Health Questionnaire Score at the End of Treatment
Description: The 28-item General Health Questionnaire is a self-reported questionnaire for the detection of non-psychotic mental disorders (anxiety and depression) in the community and primary care settings. A series of four subscale scores (ranging from 0 [good] to 21 [bad]) were combined to give a total score, which ranged from 0 (good) to 84 (bad). As such, a negative value indicates an improvement in score from baseline.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 79 | 75
units on a scale | -1.7 (11.58) | -3.0 (9.68)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline in the mean total 28-item General Health Questionnaire score at the end of treatment was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.647, ANCOVA; Estimated mean treatment difference = 0.72, 95% CI 2-sided [-2.38 to 3.82]

13. Secondary Outcome: Change From Baseline in the Mean Nine-hole Peg Test Score at the End of Treatment
Description: The Nine-Hole Peg Test is a board with nine holes into which subjects have to insert nine pegs and is designed to test dexterity and coordination. Scores range from 0 (good) to 60 (bad). As such a decrease in score indicates an improvement, and a negative value indicates an improvement from baseline.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 66 | 65
units on a scale | -0.47 (3.91) | 0.38 (2.33)

14. Secondary Outcome: Change From Baseline in the Mean Total Bladder Control Test Score at the End of Treatment
Description: The total bladder control test score was the sum score from fifteen questions were each scored on a 0-2 scale (one question 0-3), where 0 = good and 2/3 = bad. Ten questions were related to bladder symptoms and control and five were related to the effects on the patient's life. The summary parameters were the total score with a minumum possible score of 0 and a maximum possible score of 31. A decrease in score indicates an improvement, as such a negative value indicates an improvement in condition from baseline.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 58 | 60
units on a scale | -2.2 (4.63) | -1.7 (5.16)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline in the mean total bladder control test score at the end of treatment was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.889, ANCOVA; Estimated mean treatment difference = -0.12, 95% CI 2-sided [-1.77 to 1.54], Standard Error of Mean 0.83

15. Secondary Outcome: Change From Baseline in the Mean Tremor Activities of Daily Living Scale Score at the End of Treatment
Description: The tremor activities of daily living scale is a patient self-reported questionnaire which consists of 25 questions relating to the effect of tremors on different day-to-day activities, such as eating, drinking, threading a needle and tying a shoe. The ability to perform these tasks was scored on a scale of 0 (unable) to 3 (completely able). The summary parameter was the total score with a minimum of 0 (unable to perform tasks) and a maximum of 75 (completely able to perform tasks). As such, a positive value indicates an improvement in condition from baseline.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 40 | 40
units on a scale | -2.2 (6.53) | -1.2 (8.25)

16. Secondary Outcome: Change From Baseline in the Mean Ten-metre Mobility Score at the End of Treatment
Description: The 10 Metre Mobility Score is a four point scale assessing a subject's level of mobility. The time taken to walk ten metres was measured for the subset of subjects who were able to walk. A decrease in time indicates an improvement in condition.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: time (seconds)
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 38 | 47
time (seconds) | -2.78 (4.75) | -0.74 (7.85)

17. Secondary Outcome: Change From Baseline in the Mean Sleep Quality 100 mm Visual Analogue Scale Score at the End of Treatment
Description: Sleep quality scores were rated using a 100 mm visual analogue scale where 0 = best and 100 = worst. As such, a negative value is indicative of an improvement in score from baseline.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 79 | 77
units on a scale | -16.25 (27.96) | -10.05 (28.04)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The from baseline in the mean sleep quality 100 mm visual analogue scale score at the end of treatment was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.047, ANCOVA; Estimated mean treatment difference = -7.10, 95% CI 2-sided [-14.11 to -0.08]

18. Secondary Outcome: Change From Baseline in the Mean Sleep Amount 100 mm Visual Analogue Scale Score at the End of Treatment
Description: Sleep amount was rated using a 100 mm visual analogue scale where 0 = best and 100 = worst. As such, a negative value is indicative of an improvement in score from baseline.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 79 | 77
units on a scale | -13.55 (25.70) | -9.79 (26.18)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline in the mean sleep amount 100 mm visual analogue scale score at the end of treatment was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.198, ANCOVA; Estimated mean treatment difference = -4.53, 95% CI 2-sided [-11.45 to 2.40]

19. Secondary Outcome: Change From Baseline in the Mean Feeling Upon Wakening 100 mm Visual Analogue Scale Score at the End of Treatment
Description: as for outcome 18
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 79 | 77
units on a scale | -8.75 (28.91) | -9.04 (25.90)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The from baseline in the mean feeling upon wakening 100 mm visual analogue scale score at the end of treatment was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.717, ANCOVA; Estimated mean treatment difference = -1.36, 95% CI 2-sided [-8.80 to 6.07]

20. Secondary Outcome: Change From Baseline in the Mean Barthel Activities for Daily Living Scale Score at the End of Treatment
Description: The Barthel Index consists of 10 items that measure a person's daily functioning, specifically the activities of daily living and mobility. The items include feeding, moving from wheelchair to bed and return, grooming, transferring to and from a toilet, bathing, walking on level surface, going up and down stairs, dressing, continence of bowels and bladder. The person receives a score based on whether they have received help while doing the task. The ability to undertake the 10 different daily activities was assessed on scales of 0-1, 0-2 or 0-3, with 0 indicative of the poorest outcome and the highest possible score indicative of the best outcome. The summary parameter was the total score for each of the ten items, with a minimum possible score of 0 and a maximum possible score of 20. An increased score indicates an improvement, with a change of two or greater in the total score indicating a clinically relevant change. A positive value therefore indicates an improvement from baseline.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 78 | 77
units on a scale | -0.4 (1.81) | 0.1 (1.59)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline in the mean Barthel Activities for Daily Living scale score at the end of treatment was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.087, ANCOVA; Estimated mean treatment difference = -0.47, 95% CI 2-sided [-1.01 to 0.07]

21. Secondary Outcome: Change From Baseline in the Mean Short Orientation-Memory-Concentration Test at the End of Treatment
Description: The Short Orientation-Memory-Concentration test is a questionnaire designed to measure orientation, concentration on simple tasks and learning and recall of simple information. The test consists of six items, such as 'what year is it now?' and 'count backwards from 20 to 1'. Each item was scored between 0 (maximum number of errors) and three-10 (best score; no errors), with a point deducted for each error. The summary parameter was the total score from the sum of scores for each item, with an overall possible maximum score of 28 (no errors). Scores over 20 are considered 'normal'. As such, an increased score indicates an improvement, and a positive value indicates an improvement in score from baseline.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 78 | 76
units on a scale | -1.0 (5.02) | 0.0 (3.20)

22. Secondary Outcome: Change From Baseline in the Mean Reading Visual Acuity Test Score at the End of Treatment
Description: Assessment of reading visual acuity was made using a standard reading chart. Scores could range from 1 (good) to 20 (bad), indicating good and poor eyesight, respectively. As such, a negative value from baseline indicates an improvement in eyesight.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 75 | 72
units on a scale | 0.1 (1.99) | -0.0 (2.16)

23. Secondary Outcome: Change From Baseline in the Mean Care-Giver Strain Index Score at the End of Treatment
Description: The Caregiver Strain Index is a 13-item questionnaire designed to detect strain in those that care for subjects. Carers were asked if they found certain situations difficult (i.e. work adjustments, family adjustment, emotional adjustments, physical effort). Each question was scored zero (answered no) or one (answered yes), and was recorded for each of the 13 questions. The summary parameter was the total score, which was the sum score of the 13 questions, giving a minimum possible score of 0 (no strain) and maximum possible score of 13 (maximum possible strain). As such a negative value from baseline indicates an improvement in caregiver strain.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 25 | 18
units on a scale | -0.9 (2.53) | -0.1 (1.32)

24. Secondary Outcome: Change From Baseline in the Mean Guy's Neurological Disability Scale Score at the End of Treatment
Description: The Guy's Neurological Disability Scale has 12 separate categories which include cognition, mood, vision, speech, swallowing, upper limb function, lower limb function, bladder function, bowel function, sexual function, fatigue, and 'others'. Each category consists of a series of questions, which are scored on a 0 to 5 scale, with 0 being indicative of a better outcome and 5 being indicative of a worse outcome. The total Guy's Neurological Disability Scale score is the unweighted sum from the 12 categories with a minimum score of 0 and maximum of 60. A negative value indicates an improvement in score from baseline.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 66 | 63
units on a scale | -0.9 (6.20) | -2.7 (4.29)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline in the mean Guy's Neurological Disability Scale score at the end of treatment was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.048, ANCOVA; Estimated mean treatment difference = 1.81, 95% CI 2-sided [0.02 to 3.60]

25. Secondary Outcome: Change From Baseline in the Mean Total Adult Memory and Information Processing Battery Test Score at the End of Treatment
Description: The Adult Memory and Information Processing Battery test comprises six sub-sections which assess cognition and mental alertness. These include immediate and delayed story recall, word-list learning, copying a complex figure followed by its immediate reproduction, design learning, and information processing (parts A and B). The sum score for each section gave the total score which ranged from 1 (bad) to 105 (good). As such, a positive value indicates an improvement in score from baseline.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 73 | 70
units on a scale | 1.8 (5.15) | 2.1 (5.51)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline in the mean Atkinson Morley Information Processing Battery test score at the end of treatment was compared between treatment groups using ANCOVA with baseline primary impairment score as the covariate; Test type: Superiority or Other; p = 0.904, ANCOVA; Estimated mean treatment difference = -0.11, 95% CI 2-sided [-1.85 to 1.64]

ADVERSE EVENTS:
Time Frame: All adverse events occurring during the six-week parallel group treatment period were collected. All deaths and serious adverse events occurring within 28 days of the final dose of study medication were also collected.
Description: All adverse events occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | GW-1000-02 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/80 | 1/80
Other Adverse Events (participants affected / at risk) | 67/80 | 57/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GW-1000-02 (N=80) | Placebo (N=80)
UPPER RESPIRATORY TRACT INFECTION NOT OTHERWISE SPECIFIED (NOS) (Infections and infestations) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION NOT OTHERWISE SPECIFIED (Infections and infestations) | 0 | 1
SEPSIS NOS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION NOS (Infections and infestations) | 0 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
APPENDICITIS (Gastrointestinal disorders) | 0 | 1
ARTHRITIS NOS (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GW-1000-02 (N=80) | Placebo (N=80)
Dizziness (Nervous system disorders) | 25 | 10
Disturbance in attention (Nervous system disorders) | 7 | 0
Headache NOS (Nervous system disorders) | 7 | 13
Somnolence (Nervous system disorders) | 7 | 0
Oral pain (Gastrointestinal disorders) | 8 | 4
Nausea (Gastrointestinal disorders) | 7 | 5
Oral discomfort (Gastrointestinal disorders) | 7 | 7
Diarrhoea NOS (Gastrointestinal disorders) | 6 | 0
Mouth Ulceration (Gastrointestinal disorders) | 4 | 0
Fatigue (General disorders) | 12 | 3
Application site pain (General disorders) | 8 | 8
Feeling drunk (General disorders) | 4 | 0
Disorientation (Psychiatric disorders) | 6 | 0
Vertigo (Ear and labyrinth disorders) | 5 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 3
Application Site Reaction Not Otherwise Specified (General disorders) | 3 | 3
Dry Mouth (Gastrointestinal disorders) | 3 | 0
Euphoric Mood (Psychiatric disorders) | 3 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle Weakness Not Otherwise Specified (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in Limb (Musculoskeletal and connective tissue disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.